CLINICAL TRIAL: NCT02217605
Title: Investigating the Effects of an Oral Fructose Challenge on Hepatic ATP Reserves in Healthy Volunteers
Brief Title: 31P Magnetic Resonance Spectroscopy Fructose Study
Acronym: 31PMRS_FRU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Bawden (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Unilever R&D (Industry)
Responsible Party: Sponsor-Investigator, Stephen Bawden, CASE studentship researcher, University of Nottingham
Organization: University of Nottingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A32006_FRU
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: NAFLD; Oral Fructose Challenge; 31P MRS; Liver; Subjects
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fructose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fructose (Experimental): Oral Fructose Challenge (75 g fructose in 500 ml water) followed by 75 minutes 31P MRS
  Interventions: Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: Fructose — Oral Fructose Challenge (75 g fructose in 500 ml water) following overnight fast

SUMMARY:
The purpose of this study is to determine the effects of an oral fructose challenge on liver adenosine triphosphate (ATP) reserves using 31P magnetic resonance spectroscopy (MRS) as a potential measure measure of liver health.

DETAILED DESCRIPTION:
This study uses 31P spectra acquired from the liver in healthy subjects following a fructose drink to monitor ATP levels. This is also related to baseline BMI, liver glycogen and liver lipid levels

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18 - 30
* BMI 20 - 27 kg/m^2
* Healthy

Exclusion Criteria:

* Smokers
* Liver disease or Metabolic Disorders
* Metal implants (not suitable for MRI)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hepatic ATP reserves following an oral fructose challenge | 2 hours post prandial
  Monitor hepatic ATP levels following an oral fructose challenge using 31P magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Correlate hepatic ATP depletion / recovery with BMI, liver lipids and liver glycogen | 2 hours post prandial
  Measure baseline liver lipid and glycogen using magnetic resonance spectroscopy and correlate BMI, lipid and glycogen levels with rate of ATP depletion and recovery following an oral fructose challenge

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marciani, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom